CLINICAL TRIAL: NCT02659501
Title: Liposomal Bupivacaine in Implant Based Breast Reconstruction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Subhas Gupta, MD, PhD, Principal Investigator, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5150012
Record Dates: First submitted 2015-06-29; First posted 2016-01-20 (Estimated); Results first posted 2019-08-21 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2020-12

CONDITIONS: Breast Cancer; Postoperative Pain
Keywords: Breast reconstruction; Bupivacaine; Liposomal bupivacaine; Postoperative analgesia
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative | interventions — Bupivacaine; Epinephrine; Morphine; oxycodone-acetaminophen; Diazepam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bupivacaine with epinephrine injections (Active Comparator): Patients in the control arm of the study will be treated intra-operatively with standard of care, 0.5% bupivacaine and epinephrine injection (1:200,000), with 50 mg delivered into each breast pocket to perform a field block of the breast pocket (see below). Postoperatively, these patients will be treated with standard postoperative pain control, including narcotics as needed, such as morphine sulfate and hydrocodone/acetaminophen, and muscle relaxants, such as diazepam.
  Interventions: Drug: Bupivacaine with epinephrine; Drug: Morphine sulfate; Drug: Hydrocodone/acetaminophen; Drug: Diazepam
- Liposomal bupivacaine (Experimental): Patients in the experimental arm of the study will be treated intra-operatively with 1.33% liposomal bupivacaine, with 133 mg delivered to perform a field block of each breast pocket. Postoperatively, these patients will be treated with standard postoperative pain control, including narcotics as needed, such as morphine sulfate and hydrocodone/acetaminophen, and muscle relaxants, such as diazepam.
  Interventions: Drug: Liposomal bupivacaine; Drug: Morphine sulfate; Drug: Hydrocodone/acetaminophen; Drug: Diazepam

INTERVENTIONS:
Drug: Liposomal bupivacaine — Liposomal Bupivacaine is an aqueous suspension of multivesicular liposomes containing bupivacaine. After injection into soft tissue, bupivacaine is slowly released from the multivesicular liposomes, extending this drug's duration of action.
  Other Names: Exparel
  Arms: Liposomal bupivacaine
Drug: Bupivacaine with epinephrine — Bupivacaine, like other local anesthetics reduces the flow of sodium in and out of nerves. This decreases the initiation and transfer of nerve signals in the area in which the drug is injected. This leads first to a loss of sensation of pain, temperature, touch, and deep pressure. This drug is the current standard of care for local, postoperative local anesthesia following breast reconstruction. Epinephrine, a vasoconstrictor, is included in bupivacaine formulations to improve the duration of local anesthesia.
  Other Names: Marcaine; Sensorcaine
  Arms: Bupivacaine with epinephrine injections
Drug: Morphine sulfate — Morphine is an opiate pain medication administered intravenously for severe, breakthrough post-operative pain.
  Other Names: Roxanol
Drug: Hydrocodone/acetaminophen — Hydrocodone acetaminophen is a combination of an opiate pain medication (hydrocodone) and a non-steroidal anti-inflammatory drug (acetaminophen) given orally to patients for moderate post-operative pain.
  Other Names: Norco
Drug: Diazepam — Diazepam is a benzodiazepine medication that is administered orally to treat muscle spasms in patient's following expander and implant-based breast reconstruction.
  Other Names: Valium

SUMMARY:
Objectives:

1. To evaluate the effect of liposomal bupivacaine on postoperative pain levels.
2. To evaluate the effect of liposomal bupivacaine on postoperative opioid consumption and opioid related adverse events.
3. To evaluate the effect of liposomal bupivacaine on length of hospital stay.
4. To evaluate the effect of liposomal bupivacaine on patient satisfaction with postoperative pain control.
5. To evaluate the effect of liposomal bupivacaine on overall patient satisfaction.

DETAILED DESCRIPTION:
Objectives:

1. To evaluate the effect of liposomal bupivacaine on postoperative pain levels.
2. To evaluate the effect of liposomal bupivacaine on postoperative opioid consumption and opioid related adverse events.
3. To evaluate the effect of liposomal bupivacaine on length of hospital stay.
4. To evaluate the effect of liposomal bupivacaine on patient satisfaction with postoperative pain control.
5. To evaluate the effect of liposomal bupivacaine on overall patient satisfaction.

The objective of this project is to evaluate the role of liposomal bupivacaine in postoperative pain control following tissue expander and implant based breast reconstruction. This unique formulation of bupivacaine lends this drug a longer duration of action and reduced plasma bupivacaine concentrations compared to plain bupivacaine. This agent has been demonstrated to be safe, well tolerated, and effective in a number of different clinical applications. However, its role has yet to be evaluated in the context of breast reconstruction.

Thus, the authors propose the first, randomized, controlled clinical trial of liposomal bupivacaine for postoperative pain management following tissue expander and implant based breast reconstruction. Patients will be stratified into two study groups. Patients in the Group 1 (Bupivacaine) will be treated intraoperatively with injections of 0.5% bupivacaine and epinephrine 1:200,000, with 50 mg delivered to perform a field block of each pocket. This is the current standard of care. Patients in the Group 2 (Liposomal Bupivacaine) will be treated intraoperatively with injections of 1.33% liposomal bupivacaine, with 133 mg delivered to perform a field block of each breast pocket. This is the experimental intervention. Postoperatively, the investigators will assess pain levels, opioid consumption, opioid related adverse events, length of stay, and satisfaction.

The findings from this study will allow the authors to better elucidate the role of liposomal bupivacaine in expander/implant based breast reconstruction. In doing so, they may allow the authors to identify the ideal pain regimen for these patients. This holds important implications, with the potential to reduce postoperative pain, opioid consumption, opioid related adverse events, length of stay, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing immediate unilateral or bilateral tissue-expander breast reconstruction following skin-sparing or nipple-sparing mastectomy

Exclusion Criteria:

* Women who are unable to give informed consent to participate in this study
* Women with a documented history of hypersensitivity reactions to local-anesthetic agents
* Women with a diagnosis of chronic pain disorders such as fibromyalgia, chronic migraine headaches, or psychiatric disorders other than depression or anxiety
* Women who are currently pregnant
* Women undergoing tissue expander based breast reconstruction with a muscle flap in combination with a tissue expander
* Women with impaired hepatic function

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Subhas C. Gupta, MD, PhD, Principal Investigator — Loma Linda University; Wendy W. Wong, MD, Study Director — Loma Linda University
Locations (1):
- Loma Linda University Health System, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heller L, Kowalski AM, Wei C, Butler CE. Prospective, randomized, double-blind trial of local anesthetic infusion and intravenous narcotic patient-controlled anesthesia pump for pain management after free TRAM flap breast reconstruction. Plast Reconstr Surg. 2008 Oct;122(4):1010-1018. doi: 10.1097/PRS.0b013e3181858c09. PMID 18827631
- [Background] Wheble GA, Tan EK, Turner M, Durrant CA, Heppell S. Surgeon-administered, intra-operative transversus abdominis plane block in autologous breast reconstruction: a UK hospital experience. J Plast Reconstr Aesthet Surg. 2013 Dec;66(12):1665-70. doi: 10.1016/j.bjps.2013.07.017. Epub 2013 Jul 31. PMID 23910912
- [Background] Dasta J, Ramamoorthy S, Patou G, Sinatra R. Bupivacaine liposome injectable suspension compared with bupivacaine HCl for the reduction of opioid burden in the postsurgical setting. Curr Med Res Opin. 2012 Oct;28(10):1609-15. doi: 10.1185/03007995.2012.721760. Epub 2012 Sep 3. PMID 22900785
- [Background] Richard BM, Ott LR, Haan D, Brubaker AN, Cole PI, Nelson KG, Ross PE, Rebelatto MC, Newton PE. The safety and tolerability evaluation of DepoFoam bupivacaine (bupivacaine extended-release liposome injection) administered by incision wound infiltration in rabbits and dogs. Expert Opin Investig Drugs. 2011 Oct;20(10):1327-41. doi: 10.1517/13543784.2011.611499. Epub 2011 Aug 26. PMID 21867476
- [Background] Davidson EM, Barenholz Y, Cohen R, Haroutiunian S, Kagan L, Ginosar Y. High-dose bupivacaine remotely loaded into multivesicular liposomes demonstrates slow drug release without systemic toxic plasma concentrations after subcutaneous administration in humans. Anesth Analg. 2010 Apr 1;110(4):1018-23. doi: 10.1213/ANE.0b013e3181d26d2a. PMID 20357145

RESULTS

PARTICIPANT FLOW:
Groups:
- Bupivacaine With Epinephrine Injections: Patients in the control arm will be treated intra-operatively with standard of care, 0.25% bupivacaine and epinephrine injection (1:200,000), with 50 mg delivered to each breast pocket. Postoperatively, pain will be treated with narcotics as needed, such as morphine sulfate and hydrocodone/acetaminophen, and muscle relaxants, such as diazepam.
  Bupivacaine with epinephrine: Bupivacaine is a local anesthetic. This drug is the current standard of care for local anesthesia following breast reconstruction.
  Morphine sulfate: Morphine is an opiate pain medication administered intravenously for severe post-operative pain.
  Hydrocodone/acetaminophen: Hydrocodone acetaminophen is a combination of an opiate (hydrocodone) and a non-steroidal anti-inflammatory drug (acetaminophen) given orally to patients for moderate post-operative pain.
  Diazepam: Diazepam is a benzodiazepine medication that is administered orally to treat muscle spasms.
- Liposomal Bupivacaine: Patients in the experimental arm of the study will be treated intra-operatively with 1.33% liposomal bupivacaine, with 133 mg delivered to each breast pocket. Postoperatively, pain will be treated with narcotics as needed, such as morphine sulfate and hydrocodone/acetaminophen, and muscle relaxants, such as diazepam.
  Liposomal bupivacaine: Liposomal Bupivacaine is a suspension of multivesicular liposomes containing bupivacaine. After injection, bupivacaine is slowly released from the liposomes, extending this drug's duration of action.
  Morphine sulfate: Morphine is an opiate pain medication administered intravenously for severe post-operative pain.
  Hydrocodone/acetaminophen: Hydrocodone acetaminophen is a combination of an opiate (hydrocodone) and a non-steroidal anti-inflammatory drug (acetaminophen) given orally to patients for moderate post-operative pain.
  Diazepam: Diazepam is a benzodiazepine medication that is administered orally to treat muscle spasms.
Period: Overall Study
Arm/Group | Bupivacaine With Epinephrine Injections | Liposomal Bupivacaine
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine With Epinephrine Injections | Liposomal Bupivacaine | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 10 | 19
  >=65 years | 3 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (12.6) | 48.7 (11.1) | 52.4 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: The Effect of Liposomal Bupivacaine on Average Postoperative Pain Levels on Postoperative Day 1.
Description: Postoperative pain levels were determined with a numeric rating scale (NRS), rating pain from 0 - 10, where 0 = no pain, 10 = worst possible pain. Higher scores indicate a worse outcome. Pain levels were determined during routine vital signs every 4 hours post-operatively.
Time Frame: Average Pain Scores 24 hours Post-Operatively
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bupivacaine With Epinephrine Injections | Liposomal Bupivacaine
Number analyzed (Participants) | 12 | 12
score on a scale | 3.66 (0.33) | 3.68 (1.35)

2. Primary Outcome: The Effect of Liposomal Bupivacaine on Antiemetic Consumption
Description: The effect of liposomal bupivacaine on antiemetic consumption was assessed in mg of ondansetron consumed over first 24 hours post-operatively.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: mg of ondansetron
Arm/Group | Bupivacaine With Epinephrine Injections | Liposomal Bupivacaine
Number analyzed (Participants) | 12 | 12
mg of ondansetron | 7.33 (6.57) | 5.75 (4.94)

3. Primary Outcome: The Effect of Liposomal Bupivacaine on Postoperative Opioid Consumption
Description: Postoperative opioid consumption will be determined in each group. Opioid consumption post-operatively will be determined for patients in each group in standardized units of morphine milligram dosing equivalents per hour.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: Morphine equivalent dosage per hour
Arm/Group | Bupivacaine With Epinephrine Injections | Liposomal Bupivacaine
Number analyzed (Participants) | 12 | 12
Morphine equivalent dosage per hour | 1.31 (.72) | .76 (.55)

4. Primary Outcome: The Effect of Liposomal Bupivacaine on Postoperative Diazepam Consumption
Description: Benzodiazepine consumption, in mg of diazepam, was recorded for all patients and compared over the first 24 hours post-operatively.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: mg of diazepam/hr
Arm/Group | Bupivacaine With Epinephrine Injections | Liposomal Bupivacaine
Number analyzed (Participants) | 12 | 12
mg of diazepam/hr | 0.35 (0.19) | 0.18 (0.21)

5. Primary Outcome: The Effect of Liposomal Bupivacaine on Length of Hospital Stay
Description: Length of hospital stay will be determined for patients in each group, in total hours.
Time Frame: 24-60 hours
Measure: Mean (Standard Deviation); unit: hrs
Arm/Group | Bupivacaine With Epinephrine Injections | Liposomal Bupivacaine
Number analyzed (Participants) | 12 | 12
hrs | 46.7 (21.1) | 29.8 (15.3)

ADVERSE EVENTS:
Arm/Group | Bupivacaine With Epinephrine Injections | Liposomal Bupivacaine
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

LIMITATIONS AND CAVEATS:
Our trial was terminated after 12 months at 24 patients. Early termination lead to smaller numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No